CLINICAL TRIAL: NCT00183196
Title: Gabapentin as an Adjunct to Naltrexone for Alcoholism
Brief Title: Effectiveness of Gabapentin When Used With Naltrexone to Treat Alcohol Dependence Compared to Placebo and Naltrexone Alone
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Raymond F. Anton, Distinguished University Professor, Medical University of South Carolina
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NIAAAANT09568-2005a; 5R01AA009568-14 (NIH); NIH RO1 AA09568
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Results first posted 2013-05-30 (Estimated); Last update posted 2018-06-07 (Actual); Status verified 2018-05

CONDITIONS: Alcohol Dependence
Keywords: Alcohol dependence; Alcoholism; Heavy drinking
MeSH Terms: conditions — Alcoholism | interventions — Naltrexone; Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): Naltrexone plus placebo
  Interventions: Drug: Naltrexone
- 2 (Active Comparator): naltrexone + gabapentin
  Interventions: Drug: Naltrexone plus Gabapentin
- 3 (Sham Comparator): Placebo plus placebo
  Interventions: Other: Inactive Placebo

INTERVENTIONS:
Drug: Naltrexone — Naltrexone (50 mg/day) plus gabapentin placebo in divided doses for the first 6weeks. Naltrexone (50 mg/day) for rest of 16-weeks
  Arms: 1
Drug: Naltrexone plus Gabapentin — naltrexone (50 mg/day) for 16-weeks plus gabapentin (up to 1200 mg/day in divided doses) for the first 6 weeks
  Arms: 2
Other: Inactive Placebo — Placebo
  Arms: 3

SUMMARY:
The purpose of this study is to determine whether, after a period of abstinence, adding 6 weeks of gabapentin (a medication approved to treat seizures) to a standard 16-week naltrexone (an opiate blocking agent approved for the treatment of alcohol dependence) treatment protocol is helpful in decreasing relapse to drinking compared to naltrexone alone or placebo. All participants will receive alcohol counseling.

DETAILED DESCRIPTION:
Subjects will enter the trial after maintaining 4 days of abstinence. During this period multiple assessments will be collected. After entering the double blind treatment portion of the study, they will be evaluated weekly for the first month, then bi-weekly until week 12 and again at week 16. There will be two follow-up visits at weeks 28 and 40. Urinary riboflavin and pill counts will be utilized to determine compliance with the medication regime.

Comparison(s): Naltrexone (50 mg/day) alone for 16-weeks; naltrexone (50 mg/day) for 16-weeks plus gabapentin (up to 1200 mg/day in divided doses) for the first 6 weeks, or inactive placebos. All subjects will receive up to 20 sessions of individual alcohol counseling.

ELIGIBILITY:
Inclusion Criteria:

* Meet criteria for primary alcohol dependence including loss of control of drinking
* No more than one previous inpatient medical detoxification
* Consumes on average 5 standard drinks for men and 4 standard drinks for women
* Able to maintain sobriety for 4 days (with or without detox medications).
* Able to read and understand questionnaires and Informed Consent
* Lives within 50 miles of the study site

Exclusion Criteria:

* Currently meets DSM-IV criteria for any other psychoactive substance dependency disorder except nicotine dependence
* Ever abused opiates
* Any psychoactive substance abuse, except marijuana and nicotine within the last 30 days as evidenced by subject report, collateral report, or urine drug screen.
* Meets DSM-IV criteria for current Axis I disorder of major depression, panic disorder, obsessive-compulsive disorder, post-traumatic stress syndrome, bipolar affective disorder, dissociative disorder or eating disorder, schizophrenia, or any other psychotic disorder or organic mental disorder.
* Has current suicidal or homicidal ideation
* Need for maintenance or acute treatment with any psychoactive medication including antiseizure medications.
* Current use of disulfiram.
* Clinically significant medical problems, such as cardiovascular, renal, GI or endocrine problem that would impair participation or limit medication ingestion.
* Hepatocellular disease indicated by elevations of SGPT (ALT) and SGOT (AST) of at least 3.0 times normal at screening and/or after 5 days of abstinence.
* Sexually active females of child bearing potential who are pregnant (by urine HCG), nursing or who are not using a reliable form of birth control.
* Has current charges pending for a violent crime (not including DUI related offenses).
* Does not have a stable living situation and a reliable source of collateral reporting.
* Has taken an opiate antagonist drug in the last month.
* Has taken gabapentin in the last month or has experienced adverse effects from it at any time in the past.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2003-01; Primary Completion 2008-12 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond F. Anton, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Center for Drug and Alcohol Programs, Charleston, South Carolina, United States

REFERENCES:
- [Result] Anton RF, Myrick H, Wright TM, Latham PK, Baros AM, Waid LR, Randall PK. Gabapentin combined with naltrexone for the treatment of alcohol dependence. Am J Psychiatry. 2011 Jul;168(7):709-17. doi: 10.1176/appi.ajp.2011.10101436. Epub 2011 Mar 31. PMID 21454917

RESULTS

PARTICIPANT FLOW:
Groups:
- Naltrexone Plus Gabapentin and CBI: Naltrexone plus gabapentin and CBI individual counseling for 6 weeks then naltrexone and CBI for 10 additional weeks.
- Naltrexone Plus Placebo and CBI: Naltrexone plus placebo and CBI individual counseling for 6 weeks then naltrexone and CBI counseling for 10 weeks.
- Placebo Plus Placebo Plus CBI: Placebo plus placebo for 6 weeks and CBI individual counseling then placebo and CBI counseling for 10 additional weeks.
Period: Overall Study
Arm/Group | Naltrexone Plus Gabapentin and CBI | Naltrexone Plus Placebo and CBI | Placebo Plus Placebo Plus CBI
Started | 50 (2 subjects had no post-randomization data) | 50 (1 subject had no post-randomization data) | 50 (1 subject had no post-randomization data)
Completed | 30 | 35 | 32
Not Completed | 20 | 15 | 18
Not completed — Withdrawal by Subject | 18 | 11 | 13
Not completed — Adverse Event | 1 | 2 | 2
Not completed — Legal event | 1 | 1 | 1
Not completed — Required more intensive care | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Naltrexone Plus Gabapentin and CBI | Naltrexone Plus Placebo and CBI | Placebo Plus Placebo Plus CBI | Total
Number analyzed (Participants) | 50 | 50 | 50 | 150
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 50 | 49 | 49 | 148
  >=65 years | 0 | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 43 (9.8) | 44.4 (10.1) | 46.6 (9.0) | 44.6 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 10 | 31
  Male | 40 | 39 | 40 | 119
Region of Enrollment [Number; unit: participants]
  United States | 50 | 50 | 50 | 150

OUTCOME MEASURES:

1. Primary Outcome: Time to Relapse to Drinking
Description: Time to relapse drinking which is 5 standard drinks perday for males and 4 standard drinks per day for females. Subjects had a minimum of 4 days of abstinence prior to being entered into the protocol.
Time Frame: 16 weeks
Population: Subjects who entered the analysis were all people with any drinking data post randomization. There was 2 people in naltrexone plus gabapentin, 1 person in naltrexone alone and 1 person in placebo group that had no post-randomization drinking data and were therefore not included in the intent to treat analysis presented.
Measure: Mean (Standard Error); unit: days
Arm/Group | Naltrexone Plus Gabapentin and CBI | Naltrexone Plus Placebo and CBI | Placebo Plus Placebo Plus CBI
Number analyzed (Participants) | 48 | 49 | 49
days | 69.9 (6.5) | 59.6 (7.6) | 57.3 (6.7)
Statistical Analysis 1: Comparison: Naltrexone Plus Gabapentin and CBI vs Naltrexone Plus Placebo and CBI vs Placebo Plus Placebo Plus CBI; Test type: Superiority or Other; Regression, Cox; Hazard Ratio (HR) = .529, 95% CI 2-sided [.281 to .997], Standard Error of Mean 4.0
Statistical Analysis 2: Comparison: Naltrexone Plus Gabapentin and CBI vs Naltrexone Plus Placebo and CBI vs Placebo Plus Placebo Plus CBI; Test type: Superiority; p = 0.04, Regression, Cox; percent heavy drinking days at baseline was used as a covariate in the analysis as it was a predictor of overall survival independent of group

ADVERSE EVENTS:
Arm/Group | Naltrexone Plus Gabapentin and CBI | Naltrexone Plus Placebo and CBI | Placebo Plus Placebo Plus CBI
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 39/50 | 29/50 | 31/50
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Naltrexone Plus Gabapentin and CBI (N=50) | Naltrexone Plus Placebo and CBI (N=50) | Placebo Plus Placebo Plus CBI (N=50)
Dizziness (Nervous system disorders) | 20 (33) | 11 (14) | 11 (21)
somnolence (General disorders) | 39 (106) | 29 (81) | 31 (90)
Blurred vision (Eye disorders) | 16 (41) | 13 (18) | 7 (25)
Premature ejaculation (Renal and urinary disorders) | 11/39 (16) | 4/40 (4) | 8/40 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No